CLINICAL TRIAL: NCT05869981
Title: Association Between Periodontal Status and Mental Health in Postpartum Women: A Cross Sectional Study
Brief Title: Association Between Periodontal Status and Mental Health in Postpartum Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: DeeptiPerio23
Record Dates: First submitted 2023-05-05; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Mental Health Issue; Periodontitis; Periodontal Diseases
MeSH Terms: conditions — Periodontitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum women: Postpartum women (6-8 weeks to 6 months after delivery) Age 25-35 years

SUMMARY:
Background- In developing countries like India, seeking mental health care is still a taboo, and a lot of stigma is attached to consulting a psychiatric specialist or a counselor. This problem magnifies during postpartum period characterized by depressive symptoms in mothers indicating persistent low mood and feeling of worthlessness with easy fatigability, poor appetite, and sleep deprivation which leads to lack of interest in daily activities including oral health care.

Rationale- Many studies have evaluated the periodontal status during pregnancy and its consequences but only few studies have been conducted evaluating the periodontal status during the postpartum period. None of the study has evaluated the association of Mental health and periodontitis during postpartum period.

Objectives-To assess the Association between Periodontal status and Mental health in Postpartum women Methods- Periodontal Status and Mental health status (by Mental Health Inventory) will be assessed in Women during postpartum period (6-8 weeks- 6 months after delivery).

Expected outcomes- Study of periodontal status during postpartum period may contribute in elucidating this interrelationship and helps to design better prevention strategies for women's mental health.

DETAILED DESCRIPTION:
AIM To assess the Association between Periodontal status and Mental health in Postpartum women OBJECTIVES Primary objectives :- Evaluation of periodontal status and mental health status in postpartum women.

Secondary objectives:- Assessment of corelation of sociodemographic characteristics with periodontal parameters and mental health status in the postpartum women.

MATERIAL AND METHODS STUDY DESIGN AND SETTINGS The present cross sectional study will be conducted in the department of Periodontology, PGIDS, Rohtak This will be an observational cross sectional study.

STUDY PERIOD : 4 MONTHS

SAMPLE SIZE- A sample size of total 128 participants was calculated by using formula of sample size calculation with an moderate effect size 0.5 alpha =0.05 and power=0.80. n, required for each group is given by:- n=(Zα/2+Zβ)2 α2/ 2 The cross sectional study will include Women (Age 25-35 years) screened 6-8 weeks- 6 months after delivery.

METHOD OF RECRUITMENT Patients will be recruited from the Outpatient Department of Oral Medicine and Radiology, Post Graduate Institute of Medical Sciences, Rohtak.

QUESTIONNAIRE A structured questionnaire will be used to collect the socio-demographic variables, psychiatric history, interpersonal relationship, life events, and obstetric risks For Mental health assessment, a standard 38 items Mental Health Inventory (MHI)30 developed by Veit and Ware(1983) to assess the overall mental health status will be used.

MHI-38 includes 38 items divided into six subscales, consisting of two general scales,

* Psychological distress with 24 items (anxiety - 9 items, depression - 4 items, loss of behavioural/ emotional control - 9 items) and
* Psychological well-being with 14 items (overall positive affect - 10 items, emotional ties - 2 items and satisfaction with life - 1 item).

Possible answers included 1 - all of the time, 2 - most of the time, 3 - a good bit of the time, 4 - some of the time, 5 - a little of the time, 6 - none of the time. All subscales are scored so higher scores indicate more of the construct named by the subscale label. Thus, higher scores on three subscales indicate positive states of mental health and higher scores on the other three subscales indicate negative states of mental health.

Results on the scale Psychological Distress range theoretically from min. 24 to max. 142 and on the scale Psychological Well-being results theoretically range from min 14 to max.84. Higher scores on Psychological Distress indicate negative states of mind, while higher scores on Psychological Well-being indicate positive states. The overall mental health index covers all the items (results theoretically range from min. 38 to max. 226) and high values imply high psychological well-being and relatively low psychological distress. Also, high values on the general scale Psychological distress imply a negative mental health status.

Socioeconomic Status will be assessed Using Modified Kuppuswamy socioeconomic scale.

PERIODONTAL PARAMETERS:- Indices will be taken at baseline. These will be:-

* Plaque index
* Gingival index
* Probing pocket depth
* Clinical attachment loss
* Bleeding on probing PLAQUE INDEX Given by Sillness & Loe (1964) Six teeth representing the six segments of the jaws will be examined: The maxillary right first molar, lateral incisor, left first bicuspid, mandibular first molar, lateral incisor, right first bicuspid. For the scoring, a mouth mirror, a probe and a light source will be used.

GINGIVAL INDEX Given by Loe & Sillness (1963) Gingiva at six teeth, representing the six segments of the jaws will be examined: The maxillary right first molar, lateral incisor, left first bicuspid, mandibular first molar, lateral incisor, right first bicuspid. For the scoring, a mouth mirror, a probe and a light source will be used on air dried teeth and gingiva.

BLEEDING ON PROBING Bleeding on probing will be recorded as 1 if it occur within 30 sec of the probing and 0 if no bleeding occurs. After adding all the scores, total score will be divided by the total no. of surfaces accessed and multiplied by 100. It will be designed as % sites with bleeding on probing.

PROBING POCKET DEPTH It will be measured as the distance from the gingival margin to the base of the pocket using the calibrated manual periodontal probe (PCP-University of North Carolina(UNC 15 )Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of the involved teeth- mesiobuccal, midbuccal, distobuccal, mesiolingual, distolingual and midlingual.

CLINICAL ATTACHMENT LEVEL:- It will be measured from cemento-enamel junction to base of the pocket. Measurements will be made at 6 sites of the involved tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, distolingual and midlingual. The mean clinical attachment loss over all examined surfaces will be calculated.

DATA MANAGEMENT AND STATISTICAL ANALYSIS Data recorded will be processed by standard statistical analysis. The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. The Chi square test will be applied to analyse categoric data. Correlation and association between predictors and dependent variables will be analysed by correlation analysis and regression analysis.

ELIGIBILITY:
Inclusion criteria:

* Postpartum women (6-8 weeks to 6 months after delivery)
* Age 25-35 years
* Having ≥20 natural teeth

Exclusion criteria:

* Systemic disease or condition that is reported to be associated with periodontal disease, including diabetes mellitus, osteoporosis, rheumatoid arthritis, chronic renal failure, cardiovascular disease and Polycystic ovary syndrome.
* History of any Mental disorder
* History of disorders as a result of psychoactive substance use or drug abuse
* Treatment with any antidepressant drug
* Non-surgical or surgical periodontal treatment within the past 6 months before inclusion into the study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self representation of Postpartum women
Study Population: The cross sectional study will include Women (Age 25-35 years) screened 6-8 weeks- 6 months after delivery.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-06-07 (Estimated); Primary Completion 2023-09-07 (Estimated); Study Completion 2023-10-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of periodontal status and mental health status | 4 months
  Periodontal parameters:- Plaque index, Gingival index, Probing pocket depth, Clinical attachment loss
  & Bleeding on probing
  Mental health Status: A standard 38 items Mental Health Inventory (MHI-38) developed by Veit and Ware(1983) . MHI-38 items divided into six subscales, consisting of two general scales,
  * Psychological distress with 24 items (anxiety - 9 items, depression - 4 items, loss of behavioural/ emotional control - 9 items) and
  * Psychological well-being with 14 items (overall positive affect - 10 items, emotional ties - 2 items and satisfaction with life - 1 item).
  Higher scores on three subscales indicate positive states of mental health and higher scores on the other three subscales indicate negative states of mental health.

SECONDARY OUTCOMES:
Correlation of sociodemographic characteristics with periodontal status(Plaque index, Gingival index, Probing pocket depth, Clinical attachment loss, Bleeding on probing) and mental health status(Mental Health Inventory [MHI] ) | 4 months
  Socioeconomic status (SES) will be assessed using Modified Kuppuswamy socioeconomic scale Score Class 26-29 Upper (I) 16-25 Upper middle (II) 11-15 Lower middle (III) 5-10 Upper lower (IV) <5 Lower (V)

CONTACTS AND LOCATIONS:
Overall Officials: Deepti Anand, MDS, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India